CLINICAL TRIAL: NCT06957314
Title: MATCHES-Novel: MAking Telehealth Delivery of Cancer Care at Home Effective and Safe for Novel Therapies: A Hospital-at-Home Model for Tarlatamab Delivery
Brief Title: A Study of Hospital-at-Home for People Receiving Tarlatamab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-077
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: Small-cell Lung Cancer; Small Cell Lung Carcinoma; Tarlatamab; Memorial Sloan Kettering Cancer Center; 25-077; extensive stage small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Participants randomized to the control group will receive tarlatamab administration as per usual care.
- Hospital-at-Home/HAH Intervention Arm (Experimental): Participants randomized to the intervention group will receive tarlatamab administration through the hospital-at-home care delivery model.
  Interventions: Other: Hospital-at-Home/HAH

INTERVENTIONS:
Other: Hospital-at-Home/HAH — After discharge, a SeniorCare community paramedic will provide a home visit to the participant's home or residence
  Arms: Hospital-at-Home/HAH Intervention Arm

SUMMARY:
The purpose of this study is to find out whether a Hospital-at-Home (HaH) program is a more efficient way to monitor people's health after receiving tarlatamab than monitoring in the hospital (inpatient).

ELIGIBILITY:
Inclusion Criteria:

Patient

* Diagnosis of extensive stage small cell lung carcinoma (ES-SCLC)
* Treatment plan of commercially available tarlatamab monotherapy as standard of care
* Patients must be 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Patients must have adequate organ and bone marrow function, defined by the following laboratory results obtained within 28 days prior to the first study treatment:

  * ANC ≥ 1000 cells/μL (without granulocyte colony stimulating factor support within 4 weeks prior to Cycle 1, Day 1)
  * Platelet count ≥50,000/μL (without transfusion within 4 weeks prior to Cycle 1, Day 1)
  * Hemoglobin ≥8.0 g/dL (without transfusion within 4 weeks prior to Cycle 1, Day 1)
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3 X upper limit of normal (ULN). Serum bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 2 x ULN may be enrolled.
  * Estimated Glomerular Filtration Rate (eGFR) ≥ 30mL/min using the CKD-EPI formula.
* The patient is willing to give and sign informed consent
* Appropriate homebound setting as defined by one of the following:

  * Lodging at MSK Residence or hotel
  * 5 New York City boroughs, lower Westchester County (northern boundary Cross County Parkway) and Nassau County (eastern boundary Wantagh State Parkway). This is based on the community paramedic (SeniorCare) 60-minute response time catchment area. If there is any uncertainty about patient residence eligibility, the Principal Investigator will decide after discussion with SeniorCare.
* Patients must be accompanied by a caregiver for the period of time the patient is enrolled in the HaH intervention. For cases where there is uncertainty, the Principal Investigator will make the final determination.

Caregiver

* Primary caregiver as identified by patient enrolled on study

Physician

* Treating physician for patient(s) enrolled on study; managing treatment plan of commercially available tarlatamab as standard of care

Exclusion Criteria:

Patient

* Patients with a documented active infection prior to starting tarlatamab. This includes grade 3 or higher viral, bacterial, or fungal infection.
* Patients with baseline dementia or cognitive barriers
* Uncontrolled arrhythmias

Caregiver

* Caregiver deemed inappropriate by treating physician

Physician

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2028-04-23 (Estimated); Study Completion 2028-04-23 (Estimated)

PRIMARY OUTCOMES:
Number of inpatient hospital days | 14 days
  Evaluate whether HaH in combination with an enhanced oncology specific telemedicine platform is efficient by quantifying inpatient hospital days during the two 7-day periods (14 days total) after the tarlatamab infusions scheduled for C1D1 and C1D8

CONTACTS AND LOCATIONS:
Overall Officials: Robert Daly, MD, MBA, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org